CLINICAL TRIAL: NCT04148807
Title: Effectiveness of a Walking Intervention on Impact Loading and Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-11-15
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Osteoarthritis, Knee; Knee Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive walking program with gait retraining (Experimental): Participant will receive 8 gait-retraining intervention sessions.
  Interventions: Behavioral: Progressive Walking with Gait Retraining
- Progressive walking program (Active Comparator): Participant receives 8 sessions of a graded walking program.
  Interventions: Behavioral: Progressive Walking Program

INTERVENTIONS:
Behavioral: Progressive Walking with Gait Retraining — A progressive walking program with gait retraining will be performed on a treadmill at self-selected comfortable walking speed wearing an inertial measurement unit (IMU) on the medial aspect of the distal tibia. The (vertical) peak positive acceleration (PPA) of the tibia is a measure of tibial shock. Subjects will be provided real-time audio feedback to reduce PPA by 20% of their average peak PPA. During retraining sessions, a faded feedback approach will be used. Feedback will be provided continuously during the first four sessions and will be faded over the last 4 sessions. Walking time will increase over the 8 sessions.
  Arms: Progressive walking program with gait retraining
Behavioral: Progressive Walking Program — A progressive walking program will also be performed on a treadmill where subjects will walk at a self-selected comfortable speed with the same walking times per session as the retraining group without any feedback or retraining cues.
  Arms: Progressive walking program

SUMMARY:
This study investigates the feasibility of a gait-retraining program for older adults with knee osteoarthritis. The study will enroll 40 participants, with 20 receiving a gait retraining intervention and 20 receiving a graded walking program without gait retraining.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a chronic condition affecting ~12% of older adults in the United States and is a leading cause of disability. Knee pain is a common clinical manifestation that leads individuals with OA to seek medical care. Current rehabilitation approaches (e.g., bracing, taping, foot orthoses, strengthening, etc.) aim to reduce knee joint loading, a well-accepted risk factor for knee OA and pain, but are not always effective. Altering gait mechanics to reduce knee loading has also been suggested. Gait retraining studies for individuals with knee OA have focused on increasing trunk lean and toe out angle to reduce the knee adduction moment (a surrogate measure of joint loading). However, these strategies create an abnormal gait pattern and may not be the best long-term solutions due to the potential injury to other joints which may limit their overall effectiveness and applicability to clinical practice. Impact loading, another mechanical factor related to knee OA, has been reduced using gait retraining strategies in runners with knee pain. It is unknown if gait retraining strategies to decrease impact loading can reduce symptoms of knee OA. Thus, the purpose of this study is to determine the feasibility of a gait retraining program focusing on decreasing impact loading in individuals with knee OA.

At baseline, following 8 intervention sessions, and at 1-month follow-up, participants will complete questionnaires, undergo three-dimensional gait analysis, and assessment of pressure pain threshold.

Note: For participants enrolled during COVID-19 outbreak, only questionnaires will be collected at follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

Subjects with a clinical definition of knee OA using NICE guidelines:

* Age ≥ 45
* Walking related joint pain in the last week that averages ≥ 4 on 11-point numeric rating scale, where 0 = no pain and 10 = worst pain possible
* History of knee pain for at least 3 months
* Morning stiffness in the morning lasting less than 30 minutes

Exclusion Criteria:

* Walk with an assistive device
* Current use of oral opiates or centrally acting pain medications
* History of lower extremity surgery
* Underwent an intra-articular knee joint injection in the past 3 months
* Suffer from inflammatory arthritis or other conditions that affect lower extremity functions
* Currently receiving treatment for their knee and unwilling to stop this treatment for the duration of the study
* Currently pregnant
* Skin allergies to adhesives

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | through study completion, an average of 2 years
  # of participants screened per month
Enrollment rate | through study completion, an average of 2 years
  # of participants enrolled per month
Retention | through study completion, an average of 2 years
  % participants that complete all study visits

SECONDARY OUTCOMES:
Withdrawals/Terminated | through study completion, an average of 2 years
  Proportion of participants who withdraw or terminated by investigators and reasons why
Adverse events (AE)/Unanticipated problems (UP) | through study completion, an average of 2 years
  Proportion of participants with AE/UP
Vertical average loading rate | Change from baseline to conclusion of intervention, an average of 1-month
  Slope of the most linear portion of the vertical ground reaction force curve, during early stance.
Vertical instantaneous loading rate | Change from baseline to conclusion of intervention, an average of 1-month
  Maximum slope of the most vertical portion of the vertical ground reaction force curve between successive data points, during early stance.
Knee Pain with Activities | Change from baseline to conclusion of intervention, an average of 1-month
  WOMAC questionnaire, pain sub scale 0-20
Knee Pain Severity | Change from baseline to conclusion of intervention, an average of 1-month
  Visual analog scale, 0-100
Pressure pain threshold | Change from baseline to conclusion of intervention, an average of 1-month
  Assessed using hand held algometer

CONTACTS AND LOCATIONS:
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Corrigan P, Davis IS, James KA, Crossley KM, Stefanik JJ. Reducing knee pain and loading with a gait retraining program for individuals with knee osteoarthritis: Protocol for a randomized feasibility trial. Osteoarthr Cartil Open. 2020 Sep 3;2(4):100097. doi: 10.1016/j.ocarto.2020.100097. eCollection 2020 Dec. PMID 36474880